CLINICAL TRIAL: NCT06629064
Title: Identifying Clinically Relevant Neural Circuit Mechanisms of Cognitive Control Training for PTSD
Brief Title: Cognitive Control Training for Extinction in PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MHBP-001-23F; 1I01CX002760 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Stress Disorders; Stress Disorders, Traumatic; Post Traumatic Stress Disorder; PTSD; Trauma and Stressor Related Disorders
Keywords: Trauma and Stressor Related Disorders; PTSD; cognitive training; working memory; Fear Extinction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial of WMT versus a Sham training
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will occur using a code corresponding to intervention arm. Participant and provider will not know the number-condition link.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Working Memory Training (Experimental): Computer-administered working memory training program. WMT is a modified working memory capacity task designed to train working memory functioning. WMT is designed to contain high interference across trials and is adaptive to performance. As participants improve working memory, the task becomes more difficult.
  Interventions: Behavioral: Working Memory Training
- Sham Training (Sham Comparator): The Sham condition requires participants to complete a similar computer task for the same length of time. The Sham Training is a modified working memory capacity task designed to place less demands on working memory.
  Interventions: Other: Sham Training

INTERVENTIONS:
Behavioral: Working Memory Training — Computer-administered working memory training program. WMT is a modified working memory capacity task designed to train working memory functioning. WMT is designed to contain high interference across trials and is adaptive to performance. As participants improve working memory, the task becomes more difficult.
  Other Names: WMT
  Arms: Working Memory Training
Other: Sham Training — The Sham condition requires participants to complete a similar computer task for the same length of time. The Sham Training is a modified working memory capacity task designed to place less demands on working memory.
  Other Names: Sham
  Arms: Sham Training

SUMMARY:
The proposed study will test whether a working memory training (WMT) program improves fear extinction learning and its underlying neural circuitry in Veterans with posttraumatic stress disorder (PTSD). WMT is designed to improves the ability to maintain task-relevant information in mind. The project will further validate the relationship between working memory and fear extinction using novel computational and multivariate analyses that link to specific PTSD symptoms. If WMT can enhance fear extinction learning, then WMT may be a powerful adjunctive treatment that can enhance exposure therapy outcomes or be leveraged as a stand-alone treatment. This project supports the Department of Veteran Affairs mission of developing viable targets of treatment for Veterans with PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is prevalent, debilitating, and associated with significant levels of functional impairment in Veterans seeking care at the VA. Despite evidence that current treatments for PTSD are effective, a substantial portion of individuals maintain elevated PTSD symptoms after first line treatments. Mechanistic insight and tools that improve the neurocognitive and affective mechanisms that underlie successful clinical outcomes from evidence-based psychotherapies, like prolonged exposure, are highly needed. One of the most prominent mechanisms associated with therapeutic symptom reduction in PTSD is fear extinction. Indeed, extinction learning is a key theoretical treatment target in exposure-based therapies for PTSD. Fear extinction learning is not only an emotional process, but relies on an individual's cognitive control abilities, including working memory (WM). Under a WM framework, high WM ability offers the ability of an individual to adjudicate the competition between threat and extinction memory expression as they repeatedly encounter feared cues that are no longer threatening. Consistent with this hypothesis, previous investigations show replicable findings that variation in WM ability is associated with laboratory measures of fear extinction learning. The investigators have previously shown that psychophysiological and neural measures of fear extinction is a construct malleable to treatment. In civilian populations a brief WM training (WMT) designed to boost WM was effective in reducing anxiety during a speech exposure and was is effective in enhancing behavioral and neural markers of WM ability. These findings raise the intriguing possibility for the mechanistic link between WM and extinction, and that enhancing WM ability through WMT may also improve fear extinction learning success in Veterans with PTSD.

The current proposal aims to answer these questions. In a between-group design, Veterans diagnosed with PTSD will complete 8-sessions of working memory training (WMT) or sham-training (ST) over a four-week period. At pre- and post-training, Veterans will complete a standard fear acquisition & extinction learning task in addition to tasks assaying WM capacity and cognitive control. The investigators will identify whether WMT modulates behavior, psychophysiological, and neural changes in extinction learning. The investigators will further test the conceptual link between WM and extinction in Veterans with PTSD by testing whether neural circuits associated with high WM capacity and extinction learning are linked. The project is expected to determine if a cognitive control training program targeting WM capacity shows the potential to enhance behavioral and neural markers of fear extinction, mechanisms that are clearly integral to current PTSD treatments. These aims support the VA mission of testing and evaluating innovative treatment targets for PTSD. Results will provide a mechanistic foundation for future clinical trials that test whether adding WMT prior to or in conjunction with exposure based psychotherapies will improve clinical outcomes and further clarify existing mechanistic and neurobiological models of PTSD and its treatment for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Meet current DSM-5 criteria for Posttraumatic Stress Disorder
* Are willing to attend 8 total remote sessions of working memory training over course of four weeks
* Are willing to attend MRI scans pre and post working memory training
* 4-week stability on pharmacological and psychosocial treatments

Exclusion Criteria:

* A lifetime history of psychotic disorders, lifetime history of bipolar disorder
* Past-year severe substance use and severe alcohol use disorder. Mild-to-moderate alcohol use disorder will be allowed to enhance generalizability in our sample due to the high comorbidity of alcohol use and PTSD
* History of any neurological disorder that might be associated with cognitive dysfunction (e.g., cerebrovascular accident, intracranial surgery, aneurysm, seizure disorder)
* Acute suicidality requiring immediate clinical intervention
* Moderate to severe traumatic brain injury (TBI). However, mild to moderate levels of TBI (mTBI) will be included.
* Receiving benzodiazepines or medications with anticholinergic effects that may affect fear learning measures
* Inability to safely complete fMRI session (i.e., metal in body, medical implants)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral Threat Expectancy Ratings During Extinction Performance | Baseline, Approximately 5 or 6 weeks
  Threat Expectancy Ratings. Behavioral ratings will be collected during the extinction learning task. Responses will be on scale of 1- 4. High scores reflect greater threat expectancy. It is expected that the working memory training group (WMT) will have lower threat expectancy ratings during extinction learning than the Sham group.
Extinction Electrodermal Activity Response | Baseline, Approximately 5 or 6 weeks
  Electrodermal Activity Response. Responses are measured in microsiemens and time-locked to the CS+ trials during extinction learning. It is expected that the working memory training group (WMT) will have lower electrodermal activity responses during extinction learning than the Sham group.
Extinction Blood Oxygen Level Dependent (BOLD) Response | Baseline, Approximately 5 or 6 weeks
  Functional Magnetic Resonance Imaging (fMRI) will be used to measure Blood Oxygen Level Dependent (BOLD) Response during the Extinction task. BOLD response during the extinction task conditions are measured using % signal change from baseline BOLD activity with higher scores indicating greater activation. It is expected that the working memory training group (WMT) will have greater changes in BOLD responses during extinction learning than the Sham group.

SECONDARY OUTCOMES:
Working Memory Task Blood Oxygen Level Dependent (BOLD) Response | Baseline, Approximately 5 or 6 weeks
  Functional Magnetic Resonance Imaging (fMRI) will be used to measure Blood Oxygen Level Dependent (BOLD) Response during a working memory capacity task while undergoing functional MRI. BOLD response to the task conditions is measured using % signal change with higher scores indicating greater activation.
Working memory capacity change detection task | Baseline, Approximately 5 or 6 weeks
  This behavioral task measures the number of visual items maintained in working memory and is a measure of working memory capacity. This task will use simple geometric shapes as stimuli. Scores are measured using percent accuracy (o - 100%) and a measure of working memory capacity (K-score range: 0 - 6 in this task). High scores indicate greater accuracy and working memory capacity.
Affective working memory task | Baseline, Approximately 5 or 6 weeks
  An affective working memory task. A behavioral task, the affective working memory task measures working memory capacity - how many stimuli are stored in working memory) and include conditions with an emotional distractors. Scores are measured using percent accuracy (range: 0-100%) and a measure of working memory capacity (K-score range: 0 - 2 in this task). High scores indicate greater accuracy and working memory capacity. Reaction time (in milliseconds) will also be collected. High Reaction time indicates slower or more impaired working memory ability.
Flanker Task | Baseline, Approximately 5 or 6 weeks
  This behavioral task measures cognitive and motor inhibition. Stimuli consist of arrows presented at the center of a computer screen. Reaction Time (in milliseconds) for button presses will be the primary variable. High scores indicate slower reaction time to make the required behavioral response. We will also measure accuracy, with high scores indicating higher accuracy and will be scored as percent correct (range: 0-100%)
Affective stop signal task | Baseline, Approximately 5 or 6 weeks
  This behavioral task measures cognitive and motor inhibitory control and will include affective stimuli. Primary outcome variables will be reaction time (in milliseconds) and accuracy (0 to 100%). High reaction time indicates slow inhibitory control on stop signal trials.

OTHER OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline, Approximately 5 or 6 weeks
  Self-reported Posttraumatic Stress Disorder (PTSD) symptoms will be measured using the PTSD Checklist for DSM-5 (PCL-5).The total score ranges from 0-80, with higher scores indicating higher severity.
PHQ-9 (Patient Health Questionnaire-9) | Baseline, Approximately 5 or 6 weeks
  Depression symptoms will be measured using the PHQ-9 (Patient Health Questionnaire-9). Scores range from 0 - 27. Higher scores indicating higher depression symptoms and severity.
General Anxiety Disorder 7 (GAD-7) | Baseline, Approximately 5 or 6 weeks
  Anxiety symptoms will be measured with the General Anxiety Disorder 7 (GAD-7). The total score ranges from 0-21. High scores indicate higher levels of anxiety symptoms.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline, Approximately 5 or 6 weeks
  Clinician-rated Posttraumatic Stress Disorder (PTSD) symptoms and PTSD diagnostic status will be measured using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Symptom severity ranges from 0 - 80. High scores indicate greater PTSD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Stout, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No